CLINICAL TRIAL: NCT05071027
Title: Dual Antiplatelet Therapy Adherence With Reminder App Usage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is discontinuing the study since the platform/Application is no longer available for use. Study terminated effective 7/29/2024.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-13195
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Aneurysm Cerebral (Unruptured)
Keywords: aneurysm; unruptured; antiplatelet; adherence; reminder; medication; DAPT
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Medication Reminder Group (Experimental): Patients in this group will receive dual antiplatelet medication reminders.
  Interventions: Other: Endovascular Neurosurgery
- Non-app Using Group (No Intervention): Patients in this group receive the same standard of care [i.e. endovascular stent-based treatment of unruptured aneurysms] as the other group, but do not receive app dual antiplatelet reminders.

INTERVENTIONS:
Other: Endovascular Neurosurgery — Custom Dual Antiplatelet Therapy reminders for patients receiving endovascular treatment of cerebral unruptured aneurysms. The app utilized to generate reminders is available on the Apple app store.
  Arms: App Medication Reminder Group

SUMMARY:
The purpose of this study is to evaluate Dual Antiplatelet Therapy adherence in patients undergoing stent-based endovascular treatment for unruptured cervical and intradural, intracranial aneurysms. Patients will be randomized on a 1:1 basis to either a medication reminder app group or a control group, with patients in both groups receiving the standard of care. The app in question, Endovascular Neurosurgery, is available on the app store. The app does not collect user data and has not been officially deemed HIPAA compliant. The only data inputted into the app are the patient's procedure date and the antiplatelet medications the patient has been prescribed. The app does not possess sensitive patient data. Patients will input the time notifications will be sent and the app will be available in both Spanish and English. The investigators will be assessing medication adherence via the Adherence Barriers Questionnaire.

DETAILED DESCRIPTION:
This will be a randomized control trial, with patients undergoing stent-based endovascular treatment for unruptured cervical and intradural, intracranial aneurysms. Informed consent will be obtained from participating patients. Patients will be assigned to either the app group or the control group.

The particular stent-based therapy, either flow-diverter devices (FDD) placement or stent-assisted coiling, will be chosen for each patient by the clinical team. During the study consultation, the app group will have the app installed on their smart phones and will be trained in its usage. Thromboelastography (TEG) and Aspirin inhibition percentage will be determined for each patient following the procedure. Patients with TEG less than 60% will have Dual Antiplatelet Therapy (DAPT] changed from 81 mg aspirin and 75 mg clopidogrel to 81 mg aspirin and 10 mg prasugrel. Patients with aspirin inhibition percentages of less than 20% will have their aspirin doses increased to 325 mg. Medication compliance of all participants will be assessed on the day of the procedure via a medication compliance questionnaire. The same questionnaire will be administered during follow-up appointments 2-4 weeks and 6 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must speak either English or Spanish fluently
* Physically able to come to the research site location.
* Elective stent-based procedures for unruptured cervical, and intracranial, intradural aneurysms
* Endovascular therapy must be deemed appropriate by clinical team.

Exclusion Criteria:

* Presence of aneurysm where treatment plan does not include dual anti-platelet therapy
* Presence of comorbidities that preclude the possibility of treatment.
* Presence of contraindications to Dual Antiplatelet Therapy.
* Presence of certain vessel anatomical characteristics.
* Lack of iPhone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Altschul, MD, Principal Investigator — Associate Professor in The Leo M. Davidoff Department of Neurological Surgery at Montefiore
Locations (1):
- Montefiore Medical Center Department of Neurosurgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient died prior to being administered the application. They were randomized into the "App Medication Reminder Group" but never received the application.
Period: Overall Study
Arm/Group | App Medication Reminder Group | Non-app Using Group
Started | 3 | 6
Completed | 2 | 2
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Population: The remaining of the patients did not complete the follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | App Medication Reminder Group | Non-app Using Group | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Spanish/Hispanic/Latino | 0 | 1 | 1
  Black or African-American | 2 | 1 | 3
  Spanish/Hispanic/Latino | 0 | 4 | 4
  Other, Not Spanish/Hispanic/Latino | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Medication Adherence
Description: Change in medication adherence from the day of the procedure to ultimately 6 months post-procedure, as assessed by a medication compliance score generated by the Adherence Barrier Questionnaire. This score ranges from 14 to 52 and a higher score indicates that a patient faces greater barriers to medication adherence.
Time Frame: Day of Procedure, 2-4 weeks post-procedure, 6 months post-procedure
Population: Data related to 'Change in Medication Adherence' was unable to be collected in order to obtain an Adherence Barrier Questionnaire Score and, as such, this Outcome was unable to be evaluated.
Arm/Group | App Medication Reminder Group | Non-app Using Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Dual Antiplatelet Therapy Non-adherence Associated Mortality
Description: Mortality data associated with non-adherence to Dual Antiplatelet Therapy is summarized by study arm/group.
Time Frame: Up to 6 months post-procedure
Population: Two participants in each arm/group were able to be evaluated for Dual Antiplatelet Therapy Non-adherence associated mortalities. Other participants were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | App Medication Reminder Group | Non-app Using Group
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

3. Secondary Outcome: Dual Antiplatelet Therapy Non-adherence Associated Morbidity and Related Adverse Events
Description: Instances of stroke/thrombotic events, all-cause morbidity, rehospitalization for cerebrovascular events, peri-treatment hospitalization lasting more than 15 days, and delayed discharge from hospital related to non-adherence to Dual Antiplatelet Therapy, were summarized by study arm/group.
Time Frame: Up to 6 months post-procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | App Medication Reminder Group | Non-app Using Group
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | App Medication Reminder Group | Non-app Using Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT05071027/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05071027/ICF_001.pdf